CLINICAL TRIAL: NCT01945593
Title: A Phase 3b Continuation Study of the Safety and Efficacy of PEGylated Recombinant Factor VIII (PEG-rFVIII; BAX 855) in Prophylaxis of Bleeding in Previously Treated Patients With Severe Hemophilia A
Brief Title: BAX 855 Continuation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 261302; 2013-002236-24 (EudraCT Number)
Record Dates: First submitted 2013-09-16; First posted 2013-09-18 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fixed BAX855 prophylaxis (Experimental): 45-80 IU/kg twice weekly to once per week.
  Interventions: Biological: BAX855
- Pharmacokinetic (PK)-tailored BAX 855 prophylaxis (Experimental): PK-tailored prophylactic BAX855 regimen based on participant's individual PK profile to maintain a Factor VIII (FVIII) trough level
  Interventions: Biological: BAX855

INTERVENTIONS:
Biological: BAX855 — Antihemophilic Factor (Recombinant), PEGylated
  Other Names: ADYNOVATE; BAX 855; PEGylated Recombinant Factor VIII

SUMMARY:
To continue the evaluation of the safety and efficacy of BAX 855 for prophylaxis and treatment of bleeding episodes in adult and pediatric previously treated patients (PTPs) aged ≤ 75 years of age with severe hemophilia A.

ELIGIBILITY:
INCLUSION CRITERIA

Participants Transitioning from Other BAX 855 Studies:

Participants transitioning from other BAX 855 studies can be provided with the continuation study informed consent form (ICF) prior to the end of study visit to review and consider participation in this continuation study. These participants will complete any additional screening assessments within 2 weeks of the previous study's end of study visit and will return to the study site within 6 (± 1) weeks of the previous study end of study visit to confirm eligibility for this continuation study.

* Participants transitioning from other BAX 855 studies who meet ALL of the following criteria are eligible for this study:

  1. Participant has completed a previous BAX 855 study and is willing to immediately transition into this continuation study.
  2. Participant is ≤75 years of age at screening of the previous BAX 855 study.
  3. Participant continues to have a Karnofsky (for participants aged ≥ 16 years) or Lansky (for participants aged < 16 years) performance score of ≥ 60.
  4. Participant is human immunodeficiency virus negative (HIV-); or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm^3, as confirmed by central laboratory at screening.
  5. Participant is hepatitis C virus negative (HCV-) by antibody or polymerase chain reaction (PCR) testing (if positive, antibody titer will be confirmed by PCR), as confirmed by central laboratory at screening; or HCV+ with chronic stable hepatitis.
  6. If female of childbearing potential, participant presents with a negative urine pregnancy test and agrees to employ adequate birth control measures for the duration of the study.
  7. Participant and/or legally authorized representative is willing and able to comply with the requirements of the protocol.
* BAX 855 Naïve Participants:

BAX 855 naïve participants who are ≥ 12 years of age can only be enrolled in this continuation study after enrollment in the phase 2/3 pivotal study is closed. BAX 855 naïve participants who are < 12 years of age can only be enrolled in this continuation study after enrollment in the pediatric previously treated patient (PTP) study is closed.

- Enrolment of BAX 855 naïve participants will only start once the sponsor has notified the study sites accordingly.

BAX 855 naïve participants who meet ALL of the following criteria are eligible for this study:

1. Participant is ≤75 years of age at screening.
2. Participant is naïve to BAX 855.
3. Participant has severe hemophilia A (FVIII clotting activity < 1%) as confirmed by central laboratory at screening after at least a 72-hour washout period.
4. Participant aged ≥ 6 years has documented previous treatment with plasma-derived FVIII or rFVIII for ≥ 150 exposure days (EDs).
5. Participant aged < 6 years has documented previous treatment with plasma-derived FVIII concentrates or rFVIII for ≥ 50 EDs.
6. Participant is currently receiving prophylaxis or on-demand therapy with FVIII.
7. Participant has a Karnofsky (for participants aged ≥ 16 years) or Lansky (for participants aged < 16 years) performance score of ≥ 60.
8. Participant is HIV-; or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm^3, as confirmed by central laboratory at screening.
9. Participant is HCV- by antibody or PCR testing (if positive, antibody titer will be confirmed by PCR), as confirmed by central laboratory at screening; or HCV+ with chronic stable hepatitis.
10. If female of childbearing potential, participant presents with a negative urine pregnancy test and agrees to employ adequate birth control measures for the duration of the study.
11. Participant and/or legally authorized representative is willing and able to comply with the requirements of the protocol.

EXCLUSION CRITERA

- Participants Transitioning from Other BAX 855 Studies:

Participants transitioning from other BAX 855 studies who meet ANY of the following criteria are not eligible for this study:

1. Participant had detectable factor VIII (FVIII) inhibitory antibodies (≥ 0.6 Bethesda unit (BU) using the Nijmegen modification of the Bethesda assay) as confirmed by central laboratory at screening.
2. Participant has developed FVIII inhibitory antibodies (≥ 0.6 BU using the Nijmegen modification of the Bethesda assay as determined at central laboratory in a previous BAX 855 study).
3. Participant has acquired a hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease) in a previous BAX 855 study.
4. Participant has severe chronic hepatic dysfunction (eg, ≥ 5 times upper limit of normal alanine aminotransferase [ALT], as confirmed by central laboratory at screening).
5. Participant has severe renal impairment (serum creatinine > 2.0 mg/dL), as confirmed by central laboratory at screening.
6. Participant experienced a life-threatening or gastrointestinal bleeding episode within 3 months prior to study entry.
7. Participant is scheduled to use other PEGylated drugs during study participation.
8. Participant is planning to take part in any other clinical study during the course of the continuation study, with the exception of any other parallel BAX 855 study.
9. Participant has medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant safety or compliance.
10. Participant is a family member or employee of the investigator.

    * BAX 855 Naïve Participants:

BAX 855 naïve participants who meet ANY of the following criteria are not eligible for this study:

1. Participant has detectable FVIII inhibitory antibodies (≥ 0.6 BU using the Nijmegen modification of the Bethesda assay) as confirmed by central laboratory at screening.
2. Participant has history of FVIII inhibitory antibodies (≥ 0.6 BU using the Nijmegen modification of the Bethesda assay or the Bethesda assay) at any time prior to screening.
3. Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease).
4. Participant has known hypersensitivity towards mouse or hamster proteins, polyethylene glycol (PEG), or Tween 80.
5. Participant has severe chronic hepatic dysfunction eg, ≥ 5 times upper limit of normal ALT, as confirmed by central laboratory at screening).
6. Participant has severe renal impairment (serum creatinine > 2.0 mg/dL), as confirmed by central laboratory at screening.
7. Participant experienced a life-threatening or gastrointestinal bleeding episode within 3 months prior to study entry.
8. Participant has current or recent (< 30 days) use of other PEGylated drugs prior to study participation or scheduled use of such drugs during study participation.
9. Participant has participated in another clinical study involving an IP other than BAX 855 or device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an investigational product (IP) or investigational device during the course of this study.
10. Participant has medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant safety or compliance.
11. Participant is a family member or employee of the investigator.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (89):
- United States (21):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Colorado, Aurora, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - North Shore-Long Island Jewish Health System, New Hyde Park, New York
  - New York - Presbyterian/Weill Cornell Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Penn State Hershey Cancer Center, Hershey, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - University of Utah, Salt Lake City, Utah
  - Puget Sound Blood Group, Seattle, Washington
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Austria (2):
  - Landes-Frauen-und Kinderklinik Linz, Linz
  - Universitatsklinik fur Innere Medizin I, Vienna
- Bulgaria (3):
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - SHAT of Oncohaematology Diseases, Sofia
  - MHAT 'Sv. Marina', EAD, Varna
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice v Motole, Prague
- Germany (4):
  - Werlhof-Institut GmbH, Hanover, Lower Saxony
  - Gerinnungszentrum Rhein-Ruhr, Duisburg, North Rhine-Westphalia
  - Vivantes Klinikum im Friedrichshain - Landsberger Allee, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Prince of Wales Hospital, Shatin, Hong Kong
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Chaim Sheba Medical Center, Ramat Gan
- Japan (7):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - University of Occupational and Environmental Health Hospital, Kitakyushu-shi, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - St. Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Ogikubo Hospital, Suginami City, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo-To
- Lithuania (2):
  - Vilnius University Hospital Santariskiu Clinics, Public Institution, Vilnius
  - Children's Hospital, Affiliate of Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Malaysia (6):
  - Penang General Hospital, George Town, Pulau Pinang
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Ampang, Ampang, Selangor
  - Pusat Darah Negara, Kuala Lumpur
  - Hospital Pulau Pinang, Pulau Pinang
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wojewodzki Szpital Specjalistyczny im.M.Kopernika w Lodzi, Lodz
- Sanador SRL, Bucharest, Romania
- Russia (2):
  - LLC "Alba Dent", Kirov
  - Regional Clinical Hospital, Krasnoyarsk
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Pusan National University Hospital, Busan
  - Eulji University Hospital, Daejeon
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (5):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Regional Universitario de Malaga, Málaga, Málaga
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Sjukhusapoteket Malmo, Malmo
  - Karolinska, Stockholm
- Universitaetsspital Zuerich, Zurich, Switzerland
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (3):
  - Ankara University Medical Faculty, Ankara
  - Akdeniz University Faculty of Medicine, Antalya
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
- Ukraine (2):
  - SI V.K.Gusak Emergency and Reconstructive Surgery Institute of NAMSU, Donetsk
  - SI Institute of Blood Pathology and Transfusion Medicine of NAMSU, Lviv
- United Kingdom (9):
  - Bristol Royal Hospital for Children, Bristol, Avon
  - St Thomas' Hospital, London, Greater London
  - Royal Free Hospital, London, Greater London
  - Great Ormond Street Hospital for Children, London, Greater London
  - Royal Manchester Children's Hospital, Manchester, Greater Manchester
  - Southampton General Hospital, Southampton, Hampshire
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Birmingham Children's Hospital, Birmingham, West Midlands
  - The Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 86 centers in 23 countries between 15 October 2013 (first participant first visit) and 02 March 2018 (last participant last visit).
Pre-assignment Details: A total of 218 subjects were enrolled, of them 216 subjects received treatment.
Groups:
- BAX 855: Age < 2 Years: Participants of age less than (<) 2 years received an infusion of 50 +/- 10 International Units (IU)/kilogram (kg) of BAX 855 twice weekly; could be increased to 80 IU/kg or a pharmacokinetically tailored (PK-tailored) prophylactic dose (should not exceed 80 IU/kg and the FVIII peak level was not to exceed 200%) at least twice weekly based on the participant's individual PK to maintain Factor VIII (FVIII) trough levels of greater than or equal to (>=) 3% until at least 100 exposure days (EDs) were reached.
- BAX 855: Age >= 2 to <12 Years: Participants of age >= 2 to <12 years received an infusion of 50 +/- 10 IU/kg of BAX 855 twice weekly; could be increased to 80 IU/kg or a PK-tailored prophylactic dose (should not exceed 80 IU/kg and the FVIII peak level was not to exceed 200%) at least twice weekly based on the participant's individual PK to maintain FVIII trough levels of >= 3% until at least 100 EDs were reached.
- BAX 855: Age >= 12 to <17 Years: Participants of age >= 12 to <17 years received an infusion of 45 +/- 5 IU/kg of BAX 855 twice weekly; could be increased to 80 IU/kg or a PK-tailored prophylactic dose (should not exceed 80 IU/kg and the FVIII peak level was not to exceed 200%) at least twice weekly based on the participant's individual PK to maintain FVIII trough levels of >= 3% until at least 100 EDs were reached.
- BAX 855: Age >= 17 Years: Participants of age >= 17 years received an infusion of 45 +/- 5 IU/kg of BAX 855 twice weekly; could be increased to 80 IU/kg or a PK-tailored prophylactic dose (should not exceed 80 IU/kg and the FVIII peak level was not to exceed 200%) at least twice weekly based on the participant's individual PK to maintain FVIII trough levels of >= 3% until at least 100 EDs were reached.
Period: Overall Study
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Started | 3 | 64 | 26 | 125
Completed | 3 | 56 | 23 | 105
Not Completed | 0 | 8 | 3 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 4
Not completed — Protocol Violation | 0 | 2 | 1 | 3
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Other: Terminated | 0 | 0 | 0 | 1
Not completed — Other: Surgical Procedure | 0 | 2 | 0 | 6
Not completed — Other: Screen Failure | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants with at least 1 BAX855 infusion.
Groups:
- BAX 855: Age < 2 Years: Participants of age < 2 years received an infusion of 50 +/- 10 IU/kg of BAX 855 twice weekly; could be increased to 80 IU/kg or a PK-tailored prophylactic dose (should not exceed 80 IU/kg and the FVIII peak level was not to exceed 200%) at least twice weekly based on the participant's individual PK to maintain FVIII trough levels of >= 3% until at least 100 EDs were reached.
- Total: Total of all reporting groups
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years | Total
Number analyzed (Participants) | 3 | 62 | 26 | 125 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.0 (0.00) | 6.0 (2.47) | 13.8 (1.30) | 33.5 (11.68) | 22.8 (15.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 1
  Male | 3 | 61 | 26 | 125 | 215
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 7 | 10
  Not Hispanic or Latino | 3 | 59 | 26 | 118 | 206
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 15 | 5 | 37 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 0 | 4
  White | 2 | 42 | 20 | 88 | 152
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Inhibitory Antibodies to Factor VIII (FVIII)
Description: Inhibitory antibodies to Factor VIII were measured by the Nijmegen modification of the Bethesda assay. Inhibitors had to be confirmed by 2 separate assessments within a 2 to 4 week period from the central laboratory.
Time Frame: Baseline through end of study (53 months)
Population: Safety analysis set (SAS) included all participants with at least 1 BAX 855 infusion. The analysis included participants that developed inhibitory antibodies (IA) to FVIII and participants that did not develop IA to FVIII and had 100 or more exposure days (ED) to BAX 855 across all studies and a FVIII inhibitory test result after the 100th ED.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 57 | 26 | 118
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Annualized Bleed Rate (ABR) - Spontaneous Bleeds
Description: The ABR was assessed based upon each individual bleeding episode. A bleeding episode was defined as subjective (pain consistent with a joint bleed) or objective evidence of bleeding which may or may not require treatment with FVIII. The ABR of spontaneous bleeds was reported separately for twice weekly, PK-t R, each of the every 5 days and every 7 days treatment regimens at the time of bleed.
Time Frame: Baseline through end of study (53 months)
Population: Full analysis set (FAS) included all participants with at least 1 BAX 855 infusion.
Measure: Median (95% Confidence Interval); unit: Bleeds per year
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 62 | 26 | 125
Bleeds per year
  Fixed-dose regimen (FDR): Every 5 Days: number analyzed (Participants) | 0 | 0 | 7 | 49
  Fixed-dose regimen (FDR): Every 5 Days |  |  | 1.381 [0.728 to 2.620] | 1.160 [0.727 to 1.852]
  FDR: Every 7 Days: number analyzed (Participants) | 0 | 0 | 1 | 14
  FDR: Every 7 Days |  |  | 0.669 [0.061 to 7.377] | 1.992 [0.822 to 4.827]
  FDR: Twice Weekly: number analyzed (Participants) | 3 | 59 | 20 | 104
  FDR: Twice Weekly | 0.614 [0.154 to 2.454] | 0.792 [0.518 to 1.210] | 1.439 [0.942 to 2.200] | 1.293 [0.913 to 1.832]
  PK-tailored regimen (PK-t R): number analyzed (Participants) | 0 | 10 | 4 | 11
  PK-tailored regimen (PK-t R) |  | 1.078 [0.450 to 2.581] | 1.602 [0.270 to 9.486] | 0.868 [0.365 to 2.067]

3. Secondary Outcome: Total Annualized Bleed Rate (ABR)
Description: The ABR was assessed based upon each individual bleeding episode. A bleeding episode was defined as subjective (pain consistent with a joint bleed) or objective evidence of bleeding which may or may not require treatment with FVIII. Bleeding occurring at multiple locations related to the same injury (e.g., knee and ankle bleed following a fall) was counted as a single bleeding episode. Total annualized bleed rate (spontaneous and traumatic bleeding episodes) was reported.
Time Frame: Baseline through end of study (53 months)
Population: FAS included all participants with at least 1 BAX 855 infusion.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 62 | 26 | 125
Bleeds per year | 1.855 (1.000) | 2.370 (3.027) | 3.175 (2.797) | 2.426 (3.258)

4. Secondary Outcome: Overall Hemostatic Efficacy Rating of BAX 855 for Treatment of Breakthrough Bleeding Episodes
Description: The participant or caregiver rated the overall treatment response at 24 (+/- 2) hours after the initiation of treatment using a 4-point efficacy rating scale as Excellent: Full relief of pain and cessation of objective signs of bleeding after a single infusion and no additional infusion is required for the control of bleeding; Good: Definite pain relief and/or improvement in signs of bleeding after a single infusion and possibly requires more than 1 infusion for complete resolution; Fair: Slight relief of pain and slight improvement in signs of bleeding after a single infusion and required more than 1 infusion for complete resolution and None: No improvement or condition worsens.
Time Frame: Baseline through end of study (53 months)
Population: FAS included all participants with at least 1 BAX 855 infusion. Here 'N' refers to the number of participants evaluable for this outcome.
Measure: Number; unit: Treated bleeds
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 43 | 24 | 95
Treated bleeds
  Excellent | 3 | 108 | 98 | 229
  Good | 3 | 66 | 49 | 250
  Fair | 0 | 5 | 7 | 36
  None | 0 | 0 | 1 | 3
  Not Reported | 0 | 13 | 13 | 26

5. Secondary Outcome: BAX 855 Infusions Needed to Treat Bleeding Episodes
Description: The BAX 855 infusions to treat each bleeding episode was determined by the participant, the participant's caregiver, and/or investigator, and was based upon the participant's response to treatment. A bleeding episode was defined as subjective (pain consistent with a joint bleed) or objective evidence of bleeding which may or may not require treatment with FVIII.
Time Frame: Baseline through end of study (53 months)
Population: FAS included all participants with at least 1 BAX 855 infusion.
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 62 | 26 | 125
Infusions | 1.3 (0.52) | 1.4 (1.14) | 1.4 (1.81) | 1.4 (1.10)

6. Secondary Outcome: Total Time Intervals Between Bleeding Episodes
Description: The time interval between bleeding episodes was calculated based upon the date and time reported for each bleeding episode. A bleeding episode was defined as subjective (pain consistent with a joint bleed) or objective evidence of bleeding which may or may not require treatment with FVIII.
Time Frame: Baseline through end of study (53 months)
Population: FAS included all participants with at least 1 BAX 855 infusion. Here number of participants analyzed refers to the number of participants evaluable for this outcome.
Measure: Median (Full Range); unit: Months
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 2 | 36 | 21 | 84
Months | 5.700 [4.074 to 7.327] | 5.051 [0.756 to 14.867] | 5.232 [1.228 to 14.571] | 5.818 [0.617 to 22.686]

7. Secondary Outcome: Average Dose of BAX 855 Per Prophylactic Infusion
Description: The average dose of BAX 855 per prophylactic infusion was reported.
Time Frame: Baseline through end of study (53 months)
Population: SAS included all participants with at least 1 BAX 855 infusion.
Measure: Mean (Standard Deviation); unit: International units per kilogram (IU/kg)
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 62 | 26 | 125
International units per kilogram (IU/kg) | 50.748 (11.312) | 53.855 (7.754) | 53.356 (10.344) | 49.727 (8.677)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an investigational product (IP), whether or not considered causally related to the IP. A serious adverse event (SAE) was defined as an untoward medical occurrence that at any dose met one or more of the following criteria: outcome was fatal/resulted in death; was life-threatening; required inpatient hospitalization or resulted in prolongation of an existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was a medically important event.
Time Frame: Baseline through end of study (53 months)
Population: SAS included all participants with at least 1 BAX 855 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 62 | 26 | 125
Participants
  AE | 3 | 52 | 18 | 101
  SAE | 0 | 7 | 4 | 22

9. Secondary Outcome: Change From Baseline in Body Temperature
Description: Change in body temperature at pre-infusion and post-infusion at end of the study was reported. In the below table, FDR refers to fixed dose regimen, PK-tR refers to PK tailored regimen at the time of sampling.
Time Frame: Baseline, end of study (53 months)
Population: SAS included all participants with at least 1 BAX 855 infusion. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 61 | 26 | 125
Degree celsius
  FDR: Pre-Infusion | -0.23 (0.208) | -0.05 (0.386) | -0.08 (0.409) | -0.01 (0.376)
  FDR: Post-Infusion | -0.07 (0.306) | -0.03 (0.394) | 0.03 (0.375) | -0.02 (0.395)
  PK-tR: Pre-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  PK-tR: Pre-Infusion |  | 0.28 (0.255) | -0.08 (0.189) | -0.10 (0.595)
  PK-tR: Post-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  PK-tR: Post-Infusion |  | 0.13 (0.362) | 0.03 (0.263) | 0.01 (0.593)

10. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change in pulse rate at pre-infusion and post-infusion at end of the study was reported. In the below table, FDR refers to fixed dose regimen, PK-tR refers to PK tailored regimen at the time of sampling.
Time Frame: Baseline, end of study (53 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 61 | 26 | 125
Beats per minute (beats/min)
  FDR: Pre-Infusion | -20.3 (21.22) | -0.1 (14.31) | -7.7 (9.07) | -0.4 (11.67)
  FDR: Post-Infusion | -13 (19.47) | 2.4 (16.72) | -6.2 (8.55) | -1 (10.07)
  PK-tR: Pre-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  PK-tR: Pre-Infusion |  | 0.1 (9.13) | -1.8 (13.91) | 4.0 (9.15)
  PK-tR: Post-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  PK-tR: Post-Infusion |  | -8.1 (14.94) | -4.5 (12.40) | -0.2 (7.31)

11. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Change in respiratory rate at pre-infusion and post-infusion at end of the study was reported. In the below table, FDR refers to fixed dose regimen, PK-tR refers to PK tailored regimen at the time of sampling.
Time Frame: Baseline, end of study (53 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Breaths per minute (breaths/min)
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 61 | 26 | 125
Breaths per minute (breaths/min)
  FDR: Pre-Infusion | -6.3 (4.73) | -0.8 (3.97) | -1.3 (1.67) | 0.4 (2.85)
  FDR: Post-Infusion | -6.3 (4.73) | -1.3 (3.55) | -1.5 (1.85) | 0.2 (2.88)
  PK-tR: Pre-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  PK-tR: Pre-Infusion |  | 1.5 (7.01) | -3.5 (5.74) | 0.2 (2.79)
  PK-tR: Post-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  PK-tR: Post-Infusion |  | 0.4 (5.73) | -3.3 (5.85) | 0.3 (2.55)

12. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Change in systolic and diastolic blood pressure at pre-infusion and post-infusion at end of the study were reported. In the below table, FDR refers to fixed dose regimen, PK-tR refers to PK tailored regimen at the time of sampling, SBP refers to systolic blood pressure, DBP refers to diastolic blood pressure.
Time Frame: Baseline, end of study (53 months)
Population: SAS with evaluable participants for this endpoint were analyzed. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 61 | 26 | 125
Millimeter of mercury (mmHg)
  SBP - FDR: Pre-Infusion | -2.7 (1.53) | 4.5 (11.82) | 4.0 (9.25) | 1.8 (12.87)
  SBP - FDR: Post-Infusion | -8.7 (8.50) | 3 (11.49) | 2.7 (8.65) | -1.4 (12.08)
  SBP - PK-tR: Pre-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  SBP - PK-tR: Pre-Infusion |  | 0.9 (8.04) | 3.5 (9.15) | 1.0 (14.54)
  SBP - PK-tR: Post-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  SBP - PK-tR: Post-Infusion |  | -1.8 (8.61) | 3.8 (6.4) | 4.9 (15.14)
  DBP - FDR: Pre-Infusion | 0.7 (8.02) | 1.8 (9.73) | 1.4 (9.69) | 1.8 (8.66)
  DBP - FDR: Post-Infusion | 5.3 (8.74) | 3 (9.72) | 0.3 (6.43) | 0.4 (9.21)
  DBP - PK-tR: Pre-Infusion: number analyzed (Participants) | 0 | 10 | 4 | 11
  DBP - PK-tR: Pre-Infusion |  | 2.3 (9.65) | 0.5 (10.28) | 1.5 (7.90)
  DBP - PK-tR: Post-Infusion: number analyzed (Participants) | 0 | 61 | 26 | 125
  DBP - PK-tR: Post-Infusion |  | -2.4 (6.67) | -2.3 (7.68) | -0.9 (7.93)

13. Secondary Outcome: Number of Participants With Shifts in Clinical Chemistry Laboratory Assessments.
Description: The number of participants with clinically significant shifts from "normal" "abnormal clinically significant (CS)" and "abnormal not clinically significant (abnormal NCS)" at baseline to "normal" "abnormal clinically significant (CS) and abnormal clinically significant (NCS)" at completion were reported. In the below table, FDR refers to fixed dose regimen at the time of sampling, AlA refers to alanine aminotransferase, AP refers to alkaline phosphatase, AsA refers to aspartate aminotransferase.
Time Frame: Baseline through end of study (53 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 60 | 26 | 125
Participants
  AlA- FDR: Normal to Normal | 3 | 43 | 20 | 55
  AlA- FDR: Normal to Abnormal NCS | 0 | 0 | 0 | 10
  AlA- FDR: Normal to Abnormal CS | 0 | 0 | 1 | 7
  AlA- FDR: Abnormal NCS to Normal | 0 | 0 | 0 | 6
  AlA- FDR: Abnormal NCS to Abnormal NCS | 0 | 1 | 0 | 14
  AlA- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 1
  AlA- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 2
  AlA- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 1
  AlA- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 3
  AP- FDR: Normal to Normal | 3 | 8 | 11 | 100
  AP- FDR: Normal to Abnormal NCS | 0 | 4 | 4 | 3
  AP- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 0
  AP- FDR: Abnormal NCS to Normal | 0 | 0 | 1 | 0
  AP- FDR: Abnormal NCS to Abnormal NCS | 0 | 4 | 0 | 2
  AP- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  AP- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 3
  AP- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  AP- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  AsA- FDR: Normal to Normal | 3 | 7 | 15 | 53
  AsA- FDR: Normal to Abnormal NCS | 0 | 0 | 0 | 12
  AsA- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 5
  AsA- FDR: Abnormal NCS to Normal | 0 | 0 | 0 | 5
  AsA- FDR: Abnormal NCS to Abnormal NCS | 0 | 0 | 0 | 7
  AsA- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  AsA- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 1
  AsA- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 1
  AsA- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  Bilirubin- FDR: Normal to Normal | 2 | 4 | 13 | 82
  Bilirubin- FDR: Normal to Abnormal NCS | 1 | 1 | 0 | 6
  Bilirubin- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 1
  Bilirubin- FDR: Abnormal NCS to Normal | 0 | 1 | 1 | 2
  Bilirubin- FDR: Abnormal NCS to Abnormal NCS | 0 | 1 | 0 | 4
  Bilirubin- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Bilirubin- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 0
  Bilirubin- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 1 | 0
  Bilirubin- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 1
  Glucose- FDR: Normal to Normal | 2 | 20 | 11 | 61
  Glucose- FDR: Normal to Abnormal NCS | 0 | 9 | 4 | 13
  Glucose- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 1
  Glucose- FDR: Abnormal NCS to Normal | 0 | 11 | 5 | 20
  Glucose- FDR: Abnormal NCS to Abnormal NCS | 1 | 3 | 1 | 8
  Glucose- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Glucose- FDR: Abnormal CS to Normal | 0 | 1 | 0 | 0
  Glucose- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Glucose- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 4

14. Secondary Outcome: Number of Participants With Shifts in Hematology Laboratory Assessments
Description: The number of participants with clinically significant shifts from "normal" "abnormal clinically significant (CS)" and "abnormal not clinically significant (abnormal NCS)" at baseline to "normal" "abnormal clinically significant (CS) and abnormal clinically significant (NCS)" at completion were reported. In the below table, FDR refers to fixed dose regimen, PK-tR refers to PK tailored regimen at the time of sampling, Leu refers to leukocytes, MCV refers to mean corpuscular volume, Lym/Leu refers to lymphocytes/leukocytes.
Time Frame: Baseline through end of study (53 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 60 | 26 | 125
Participants
  Eosinophils/Leu- FDR: Normal to Normal | 2 | 28 | 11 | 97
  Eosinophils/Leu- FDR: Normal to Abnormal NCS | 0 | 5 | 1 | 1
  Eosinophils/Leu- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 1
  Eosinophils/Leu- FDR: Abnormal NCS to Normal | 0 | 5 | 2 | 2
  Eosinophils/Leu- FDR: Abnormal NCS to Abnormal NCS | 1 | 5 | 6 | 1
  Eosinophils/Leu- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Eosinophils/Leu- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 1
  Eosinophils/Leu- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Eosinophils/Leu- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 1 | 0
  Erythrocytes MCV- FDR: Normal to Normal | 3 | 34 | 18 | 70
  Erythrocytes MCV- FDR: Normal to Abnormal NCS | 0 | 3 | 3 | 8
  Erythrocytes MCV- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 1
  Erythrocytes MCV- FDR: Abnormal NCS to Normal | 0 | 0 | 0 | 2
  Erythrocytes MCV- FDR: Abnormal NCS toAbnormal NCS | 0 | 4 | 0 | 7
  Erythrocytes MCV- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Erythrocytes MCV- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 1
  Erythrocytes MCV- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Erythrocytes MCV- FDR:Abnormal CS to Abnormal CS | 0 | 1 | 0 | 1
  Hematocrit- FDR: Normal to Normal | 2 | 34 | 15 | 84
  Hematocrit- FDR: Normal to Abnormal NCS | 0 | 0 | 2 | 3
  Hematocrit- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 3
  Hematocrit- FDR: Abnormal NCS to Normal | 0 | 6 | 4 | 6
  Hematocrit- FDR: Abnormal NCS to Abnormal NCS | 0 | 1 | 0 | 3
  Hematocrit- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Hematocrit- FDR: Abnormal CS to Normal | 0 | 1 | 0 | 0
  Hematocrit- FDR: Abnormal CS to Abnormal NCS | 1 | 0 | 0 | 1
  Hematocrit- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  Hemoglobin- FDR: Normal to Normal | 2 | 37 | 20 | 89
  Hemoglobin- FDR: Normal to Abnormal NCS | 0 | 1 | 0 | 4
  Hemoglobin- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 2
  Hemoglobin- FDR: Abnormal NCS to Normal | 0 | 3 | 0 | 3
  Hemoglobin- FDR: Abnormal NCS to Abnormal NCS | 0 | 1 | 1 | 3
  Hemoglobin- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 1
  Hemoglobin- FDR: Abnormal CS to Normal | 1 | 0 | 0 | 0
  Hemoglobin- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 1
  Hemoglobin- FDR: Abnormal CS to Abnormal CS | 0 | 1 | 0 | 0
  Leukocytes- FDR: Normal to Normal | 1 | 37 | 13 | 87
  Leukocytes- FDR: Normal to Abnormal NCS | 1 | 4 | 4 | 5
  Leukocytes- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 0
  Leukocytes- FDR: Abnormal NCS to Normal | 1 | 2 | 2 | 10
  Leukocytes- FDR: Abnormal NCS to Abnormal NCS | 0 | 0 | 1 | 1
  Leukocytes- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Leukocytes- FDR: Abnormal CS to Normal | 0 | 0 | 1 | 0
  Leukocytes- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Leukocytes- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  Lym/Leu- FDR: Normal to Normal | 0 | 39 | 19 | 98
  Lym/Leu- FDR: Normal to Abnormal NCS | 2 | 0 | 1 | 2
  Lym/Leu- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 0
  Lym/Leu- FDR: Abnormal NCS to Normal | 0 | 3 | 1 | 2
  Lym/Leu- FDR: Abnormal NCS to Abnormal NCS | 1 | 1 | 0 | 0
  Lym/Leu- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Lym/Leu- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 1
  Lym/Leu- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Lym/Leu- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  Platelets- FDR: Normal to Normal | 2 | 40 | 21 | 88
  Platelets- FDR: Normal to Abnormal NCS | 0 | 0 | 0 | 4
  Platelets- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 0
  Platelets- FDR: Abnormal NCS to Normal | 0 | 2 | 0 | 3
  Platelets- FDR: Abnormal NCS to Abnormal NCS | 1 | 0 | 0 | 3
  Platelets- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Platelets- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 1
  Platelets- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Platelets- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 1
  Hematocrit- PK-t R: Normal to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Normal to Normal | 0 | 4 | 3 | 10
  Hematocrit- PK-t R: Normal to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Normal to Abnormal NCS | 0 | 1 | 0 | 0
  Hematocrit- PK-t R: Normal to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Normal to Abnormal CS | 0 | 0 | 0 | 0
  Hematocrit- PK-t R: Abnormal NCS to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Abnormal NCS to Normal | 0 | 2 | 1 | 0
  Hematocrit- PK-t R: Abnormal NCS to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Abnormal NCS to Abnormal NCS | 0 | 0 | 0 | 0
  Hematocrit- PK-t R: Abnormal NCS to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Hematocrit- PK-t R: Abnormal CS to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Abnormal CS to Normal | 0 | 0 | 0 | 1
  Hematocrit- PK-t R: Abnormal CS to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Hematocrit- PK-t R: Abnormal CS to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hematocrit- PK-t R: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  Hemoglobin- PK-t R: Normal to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Normal to Normal | 0 | 7 | 4 | 11
  Hemoglobin- PK-t R: Normal to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Normal to Abnormal NCS | 0 | 0 | 0 | 0
  Hemoglobin- PK-t R: Normal to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Normal to Abnormal CS | 0 | 0 | 0 | 0
  Hemoglobin- PK-t R: Abnormal NCS to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Abnormal NCS to Normal | 0 | 0 | 0 | 0
  Hemoglobin- PK-t R: Abnormal NCS to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Abnormal NCS to Abnormal NCS | 0 | 0 | 0 | 0
  Hemoglobin- PK-t R: Abnormal NCS to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  Hemoglobin- PK-t R: Abnormal CS to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Abnormal CS to Normal | 0 | 1 | 0 | 0
  Hemoglobin- PK-t R: Abnormal CS to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Hemoglobin- PK-t R: Abnormal CS to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  Hemoglobin- PK-t R: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Shifts in Lipid Panel Assessments
Description: The number of participants with clinically significant shifts from "normal" "abnormal clinically significant (CS)" and "abnormal not clinically significant (abnormal NCS)" at baseline to "normal" "abnormal clinically significant (CS) and abnormal clinically significant (NCS)" at completion were reported.. In the below table, HDL refers to high density lipoprotein, LDL refers to low density lipoprotein, VLDL refers to very low density lipoprotein.
Time Frame: Baseline through end of study (53 months)
Population: SAS included all participants with at least 1 BAX 855 infusion.Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 60 | 26 | 125
Participants
  Cholesterol- FDR: Normal to Normal | 3 | 8 | 12 | 65
  Cholesterol- FDR: Normal to Abnormal NCS | 0 | 5 | 0 | 4
  Cholesterol- FDR: Normal to Abnormal CS | 0 | 0 | 2 | 2
  Cholesterol- FDR: Abnormal NCS to Normal | 0 | 0 | 3 | 8
  Cholesterol- FDR: Abnormal NCS to Abnormal NCS | 0 | 1 | 0 | 19
  Cholesterol- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 1
  Cholesterol- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 2
  Cholesterol- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  Cholesterol- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  HDL Cholesterol- FDR: Normal to Normal | 0 | 5 | 10 | 68
  HDL Cholesterol- FDR: Normal to Abnormal NCS | 0 | 2 | 3 | 13
  HDL Cholesterol- FDR: Normal to Abnormal CS | 0 | 0 | 2 | 3
  HDL Cholesterol- FDR: Abnormal NCS to Normal | 0 | 0 | 2 | 7
  HDL Cholesterol- FDR: Abnormal NCS to Abnormal NCS | 0 | 0 | 5 | 20
  HDL Cholesterol- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 1 | 0
  HDL Cholesterol- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 2
  HDL Cholesterol- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  HDL Cholesterol- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  LDL Cholesterol- FDR: Normal to Normal | 3 | 7 | 7 | 56
  LDL Cholesterol- FDR: Normal to Abnormal NCS | 0 | 2 | 0 | 9
  LDL Cholesterol- FDR: Normal to Abnormal CS | 0 | 0 | 2 | 3
  LDL Cholesterol- FDR: Abnormal NCS to Normal | 0 | 0 | 2 | 7
  LDL Cholesterol- FDR: Abnormal NCS to Abnormal NCS | 0 | 0 | 5 | 20
  LDL Cholesterol- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 1 | 0
  LDL Cholesterol- FDR: Abnormal CS to Normal | 0 | 0 | 0 | 2
  LDL Cholesterol- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  LDL Cholesterol- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  Triglycerides- FDR: Normal to Normal | 1 | 3 | 9 | 84
  Triglycerides- FDR: Normal to Abnormal NCS | 0 | 11 | 5 | 8
  Triglycerides- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 1
  Triglycerides- FDR: Abnormal NCS to Normal | 1 | 4 | 2 | 3
  Triglycerides- FDR: Abnormal NCS to Abnormal NCS | 1 | 7 | 2 | 3
  Triglycerides- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 2 | 2
  Triglycerides- FDR: Abnormal CS to Normal | 0 | 0 | 1 | 1
  Triglycerides- FDR: Abnormal CS to Abnormal NCS | 0 | 1 | 0 | 0
  Triglycerides- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 1
  VLDL Cholesterol- FDR: Normal to Normal | 3 | 30 | 14 | 67
  VLDL Cholesterol- FDR: Normal to Abnormal NCS | 0 | 4 | 2 | 8
  VLDL Cholesterol- FDR: Normal to Abnormal CS | 0 | 0 | 0 | 2
  VLDL Cholesterol- FDR: Abnormal NCS to Normal | 0 | 7 | 4 | 10
  VLDL Cholesterol- FDR: Abnormal NCS toAbnormal NCS | 0 | 0 | 0 | 14
  VLDL Cholesterol- FDR: Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 1
  VLDL Cholesterol- FDR: Abnormal CS to Normal | 0 | 0 | 1 | 1
  VLDL Cholesterol- FDR: Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  VLDL Cholesterol- FDR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0
  VLDL Cholesterol- PK-tR: Normal to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDL Cholesterol- PK-tR: Normal to Normal | 0 | 6 | 3 | 7
  VLDL Cholesterol- PK-tR: Normal to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDL Cholesterol- PK-tR: Normal to Abnormal NCS | 0 | 0 | 0 | 0
  VLDL Cholesterol- PK-tR: Normal to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDL Cholesterol- PK-tR: Normal to Abnormal CS | 0 | 0 | 0 | 0
  VLDL Cholesterol- PK-tR: Abnormal NCS to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDL Cholesterol- PK-tR: Abnormal NCS to Normal | 0 | 1 | 1 | 1
  VLDLCholesterol-PK-tR:Abnormal NCS to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDLCholesterol-PK-tR:Abnormal NCS to Abnormal NCS | 0 | 1 | 0 | 1
  VLDL Cholesterol-PK-tR:Abnormal NCS to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDL Cholesterol-PK-tR:Abnormal NCS to Abnormal CS | 0 | 0 | 0 | 0
  VLDL Cholesterol- PK-tR: Abnormal CS to Normal: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDL Cholesterol- PK-tR: Abnormal CS to Normal | 0 | 0 | 0 | 2
  VLDL Cholesterol-PK-tR:Abnormal CS to Abnormal NCS: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDL Cholesterol-PK-tR:Abnormal CS to Abnormal NCS | 0 | 0 | 0 | 0
  VLDL Cholesterol-PK-tR: Abnormal CS to Abnormal CS: number analyzed (Participants) | 0 | 10 | 4 | 11
  VLDL Cholesterol-PK-tR: Abnormal CS to Abnormal CS | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Binding Antibodies
Description: Binding antibodies (IgG and IgM) against FVIII, polyethylene glycol (PEG) and PEGylated FVIII (PEG-FVIII) were analyzed using enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline through end of study (53 months)
Population: SAS included all participants with at least 1 BAX 855 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 62 | 26 | 125
Participants
  IgG to FVIII | 0 | 2 | 1 | 2
  IgM to FVIII | 0 | 0 | 0 | 0
  IgG to PEG-FVIII | 1 | 3 | 0 | 4
  IgM to PEG-FVIII | 0 | 0 | 0 | 0
  IgG to PEG | 0 | 0 | 0 | 0
  IgM to PEG | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Anti-Chinese Hamster Ovary (CHO) Antibodies
Description: Testing for binding of anti-CHO protein antibodies was performed on citrate-anti-coagulated plasma using an ELISA employing polyclonal antihuman IgG antibodies.
Time Frame: Baseline through end of study (53 months)
Population: SAS included all participants with at least 1 BAX 855 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 3 | 62 | 26 | 125
Participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in Bleed Severity
Description: Hemophilia symptom (haemo-SYM) questionnaire has two subscales: pain and bleed. It was used to asses the bleed severity for participants >=18 years of age as: severity of spontaneous bleeding in my joints (unrelated to injury or activity), spontaneous bleeding in my muscles (unrelated to injury or activity), prolonged bleeding after injury in spite of treatment, intense pain because of bleeding event, joint pain due to active bleed and bleeding during personal hygiene routine, blood in my urine, nose bleeds and assigned a score of 0=Absent, 1=very mild, 2=mild, 3=moderate, 4=severe and 5=very severe. The score was determined as (mean score/5)*100 where mean score is the mean of the available results in the particular subscale. Higher scores on the Haemo-SYM indicate more severe symptoms. Therefore, negative change scores indicate that symptoms have improved. Here 'n' refers to the number of participants evaluable for this endpoint.
Time Frame: Baseline, end of study (53 months)
Population: FAS with population of age greater than or equal to 18 years were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 125
Score on a scale
  Fixed dose regimen: number analyzed (Participants) | 99
  Fixed dose regimen | -7.824 (18.514)
  PK-tailored regimen: number analyzed (Participants) | 9
  PK-tailored regimen | -16.667 (14.337)

19. Secondary Outcome: Change From Baseline in Pain Severity
Description: Hemophilia symptom (haemo-SYM) questionnaire has two subscales: pain and bleed. It was used to asses the pain severity for participants >=18 years of age as: pain because of swelling in my joints, climbing stairs, upon waking in the morning, active arthritis; constant pain, in my muscles, that needs medication; joint sensitivity to weather conditions; reduced range of joint movement, joint deformity, sleep disturbance because of pain or bleeds, blood in my urine, nose bleeds and assigned a score of 0=Absent, 1=very mild, 2=mild, 3=moderate, 4=severe and 5=very severe. The score was determined as (mean score/5)*100 where mean score is the mean of the available results in the particular subscale. Higher scores on the Haemo-SYM indicate more severe symptoms. Therefore, negative change scores indicate that symptoms have improved. Here 'n' refers to the number of participants evaluable for this endpoint.
Time Frame: Baseline, end of study (53 months)
Population: FAS with population of age greater than or equal to 18 years were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 125
Score on a scale
  Fixed dose regimen: number analyzed (Participants) | 99
  Fixed dose regimen | -1.341 (11.531)
  PK-tailored regimen: number analyzed (Participants) | 9
  PK-tailored regimen | -8.889 (20.659)

20. Secondary Outcome: Change From Baseline in Patient Reported Outcomes: Health-related Quality of Life (HRQoL): Short Form-36 (SF-36)
Description: HRQoL in participants aged >=14 years was measured using the SF-36 questionnaire. The questionnaire was divided into 8 domains and scored as: physical functioning (1=yes, limited a lot to 3=no, not limited at all), role-physical (1=all of the time to 5=none of the time), bodily pain (1=very severe to 6=none), general health (1=poor to 5=excellent), vitality (1=none of the time to 5=all of the time), social functioning (1=all of the time: to 5=none of the time), role emotional (1=all of the time to 5=none of the time) and mental health (1=all of the time to 5=none of the time). The score for each domain is then to be transformed to a 0-100 range as [(actual raw score-lowest possible raw score)/possible raw score range]*100. Positive change scores indicate improved HRQoL. in the below table 'FDR' indicates fixed dose regimen, 'PK-tr' indicates pharmacokinetically tailored regimen and 'n' refers to the number of participants evaluable for this endpoint.
Time Frame: Baseline, end of study (53 months)
Population: FAS with population of age greater than or equal to 14 years were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
Number analyzed (Participants) | 26 | 125
Score on a scale
  FDR: Physical functioning: number analyzed (Participants) | 8 | 75
  FDR: Physical functioning | 3.875 (4.912) | -0.108 (3.021)
  PK-t R: Physical functioning: number analyzed (Participants) | 2 | 11
  PK-t R: Physical functioning | 1.000 (1.414) | -0.364 (4.456)
  FDR: Role-physical: number analyzed (Participants) | 8 | 75
  FDR: Role-physical | 0.8 (4.13) | 0.4 (3.90)
  PK-t R: Role-physical: number analyzed (Participants) | 2 | 11
  PK-t R: Role-physical | 1.5 (3.54) | 1.2 (2.86)
  FDR: Bodily pain: number analyzed (Participants) | 8 | 75
  FDR: Bodily pain | 1.30 (2.530) | 0.81 (2.051)
  PK-t R: Bodily pain: number analyzed (Participants) | 2 | 11
  PK-t R: Bodily pain | -0.30 (2.687) | 0.39 (3.250)
  FDR: General health: number analyzed (Participants) | 8 | 74
  FDR: General health | 2.33 (3.533) | 0.48 (3.837)
  PK-t R: General health: number analyzed (Participants) | 2 | 11
  PK-t R: General health | 2.30 (0.424) | 1.56 (4.328)
  FDR: Vitality: number analyzed (Participants) | 8 | 74
  FDR: Vitality | -0.3 (3.20) | 0.1 (2.39)
  PK-t R: Vitality: number analyzed (Participants) | 2 | 11
  PK-t R: Vitality | 2.5 (3.54) | 0.7 (3.80)
  FDR: Social functioning: number analyzed (Participants) | 8 | 75
  FDR: Social functioning | 0.4 (1.69) | 0.0 (1.39)
  PK-t R: Social functioning: number analyzed (Participants) | 2 | 11
  PK-t R: Social functioning | 1.0 (1.41) | -1.2 (2.18)
  FDR: Role emotional: number analyzed (Participants) | 8 | 75
  FDR: Role emotional | -0.6 (2.26) | -0.4 (2.44)
  PK-t R: Role emotional: number analyzed (Participants) | 2 | 11
  PK-t R: Role emotional | 0.5 (0.71) | -1.1 (2.47)
  FDR: Mental health: number analyzed (Participants) | 8 | 74
  FDR: Mental health | -1.0 (1.93) | -0.3 (3.17)
  PK-t R: Mental health: number analyzed (Participants) | 2 | 11
  PK-t R: Mental health | 0.5 (0.71) | -0.5 (2.70)
  FDR: Physical component score: number analyzed (Participants) | 8 | 74
  FDR: Physical component score | 8.280 (12.985) | 1.986 (7.059)
  PK-t R: Physical component score: number analyzed (Participants) | 2 | 11
  PK-t R: Physical component score | 2.647 (7.990) | 3.414 (9.405)
  FDR: Mental component score: number analyzed (Participants) | 8 | 74
  FDR: Mental component score | -4.780 (6.680) | -1.501 (9.059)
  PK-t R: Mental component score: number analyzed (Participants) | 2 | 11
  PK-t R: Mental component score | 3.931 (7.769) | -4.185 (8.634)

21. Secondary Outcome: Change From Baseline in Patient Reported Outcomes: Health-related Quality of Life (HRQoL): Pediatrics Quality of Life (PedsQL) Questionnaire
Description: HRQoL in participants aged <14 years was measured using the PedsQL. It capture data for the following domains: physical functioning, emotional functioning, social functioning, school functioning, psychosocial functioning, physical health and a total score. Each question of the PedsQL was scored as Never: 100, almost never: 75, sometimes: 50, often: 25, almost always: 0. The mean of the individual question scores was calculated. Lower scores on the PedsQL indicating worse HRQoL. Here, FDR refers to fixed dose regimen, PK-t R refers to PK-tailored regimen. Here 'n' refers to the number of participants evaluable for this endpoint. Here 'n' refers to the number of participants evaluable for this endpoint.
Time Frame: Baseline, end of study (53 months)
Population: FAS with population of age less than 14 years were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years
Number analyzed (Participants) | 62 | 26
Score on a scale
  FDR: Physical functioning: number analyzed (Participants) | 41 | 3
  FDR: Physical functioning | 0.534 (17.896) | 3.125 (15.625)
  PK-t R: Physical functioning: number analyzed (Participants) | 7 | 2
  PK-t R: Physical functioning | -0.446 (12.425) | 7.813 (6.629)
  FDR: Emotional functioning: number analyzed (Participants) | 41 | 3
  FDR: Emotional functioning | -1.0 (16.93) | 8.3 (20.21)
  PK-t R: Emotional functioning: number analyzed (Participants) | 7 | 2
  PK-t R: Emotional functioning | -2.1 (11.85) | 10.0 (14.14)
  FDR: Social functioning: number analyzed (Participants) | 41 | 3
  FDR: Social functioning | -0.4 (16.22) | 8.3 (15.28)
  PK-t R: Social functioning: number analyzed (Participants) | 7 | 2
  PK-t R: Social functioning | -6.4 (19.73) | 5.0 (7.07)
  FDR: School functioning: number analyzed (Participants) | 36 | 3
  FDR: School functioning | 3.472 (24.107) | 15.000 (13.229)
  PK-t R: School functioning: number analyzed (Participants) | 6 | 2
  PK-t R: School functioning | -9.167 (16.591) | -12.500 (17.678)
  FDR: Psychosocial functioning: number analyzed (Participants) | 41 | 3
  FDR: Psychosocial functioning | 0.331 (15.283) | 10.556 (15.486)
  PK-t R: Psychosocial functioning: number analyzed (Participants) | 7 | 2
  PK-t R: Psychosocial functioning | -6.099 (13.025) | 0.833 (3.536)
  FDR: Total score: number analyzed (Participants) | 41 | 3
  FDR: Total score | 0.366 (14.811) | 7.971 (15.230)
  PK-t R: Total score: number analyzed (Participants) | 7 | 2
  PK-t R: Total score | -3.915 (12.201) | 3.261 (0.000)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 53 months
Description: Safety analysis was analyzed for the safety population (216 participants) and not for the enrolled population as in participant flow (218 participants).
Arm/Group | BAX 855: Age < 2 Years | BAX 855: Age >= 2 to <12 Years | BAX 855: Age >= 12 to <17 Years | BAX 855: Age >= 17 Years
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/62 | 1/26 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/3 | 7/62 | 4/26 | 22/125
Other Adverse Events (participants affected / at risk) | 3/3 | 40/62 | 12/26 | 62/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX 855: Age < 2 Years (N=3) | BAX 855: Age >= 2 to <12 Years (N=62) | BAX 855: Age >= 12 to <17 Years (N=26) | BAX 855: Age >= 17 Years (N=125)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX 855: Age < 2 Years (N=3) | BAX 855: Age >= 2 to <12 Years (N=62) | BAX 855: Age >= 12 to <17 Years (N=26) | BAX 855: Age >= 17 Years (N=125)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 2 (2) | 14 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (8) | 1 (1) | 7 (8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (8) | 1 (2) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 11 (15) | 0 (0) | 5 (5)
Ear infection (Infections and infestations) | 1 (4) | 4 (6) | 1 (2) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 13 (24) | 2 (5) | 25 (39)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 5 (9)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 4 (5) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 4 (4) | 3 (5) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 11 (22) | 1 (1) | 12 (13)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 4 (6)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 6 (6) | 1 (1) | 12 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 13 (17) | 0 (0) | 7 (8)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (5):
  • Study Protocol: Protocol (2013-06-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT01945593/Prot_000.pdf
  • Study Protocol: Protocol Amendment 1 (2013-10-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT01945593/Prot_001.pdf
  • Study Protocol: Protocol Amendment 4 (2014-05-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT01945593/Prot_002.pdf
  • Study Protocol: Protocol Amendment 7 (2015-03-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT01945593/Prot_003.pdf
  • Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT01945593/SAP_004.pdf